CLINICAL TRIAL: NCT00276445
Title: Alleviation of Cedar Pollen Induced Allergic Symptoms by Orally Taken Superfine Beta-1,3-Glucan - A Double-Blind Randomized Study
Brief Title: Alleviation of Cedar Pollen Induced Allergic Symptoms by Orally Taken Superfine Beta-1,3-Glucan
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Meiji University of Oriental Medicine (Other)
Collaborators: Kyoto Prefectural University of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 15-58-2; Japanese Minis. Edu. 17791261
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2004-01

CONDITIONS: Allergic Conjunctivitis
Keywords: allergy; Allergy conjunctivitis; beta-1-3glucan; Th1/Th2
MeSH Terms: conditions — Conjunctivitis, Allergic; Hypersensitivity | interventions — beta-1,3-glucan

INTERVENTIONS:
Drug: beta-1,3-glucan

SUMMARY:
Intravenous- injection of beta-1,3-glucan in human is known to induce T helper type 1 response, while oral uptake did not. It was examined whether superfine dispersed beta-1,3-glucan (SDG) contrived to absorbed by intestinal mucosa would alleviate allergic symptoms by per-oral ingestion

DETAILED DESCRIPTION:
Beta-1,3-glucan made from Japanese mushroom is commercially available for healthy foodstuffs. Allergy patients were orally administrated either SDG (n=30) or non-dispersed beta-1,3-glucan (NDG, n=30) and allergic symptoms were assessed clinically, by the double-blind, placebo-controlled, randomized study

ELIGIBILITY:
Inclusion Criteria:

* history of seasonal allergic conjunctivitis with or without rhinitis in spring (Japanese cedar pollen season) every year
* positive allergen specific IgE (> 30 IU/ml) or positive skin prick test result (wheal diameter > 3mm) to Japanese cedar, Orchard Grass pollen, or house dust-mite extract

Exclusion Criteria:

* Patients who had undergone immunotherapy in the previous 5 years
* a history of other immunological or medically relevant diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-01; Study Completion 2004-06

PRIMARY OUTCOMES:
Symptoms were assessed clinically by score on a allergic symptom rating scale.

SECONDARY OUTCOMES:
Total IgE and allergen specific IgE were measured.
The binding capacity of beta-1,3-glucan to peripheral CD14+ cells were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yamada, M.D. Ph.D., Principal Investigator — Meiji University of Oriental Medicine; Junji Hamuro, Ph.D., Study Director — Kyoto Prefectural University of Medicine; Shigeru Kinoshita, M.D. Ph.D., Study Chair — Kyoto Prefectural University of Medicine
Locations (1):
- Meiji University of Oriental Medicine, Kyoto, Kyoto, Japan

REFERENCES:
- [Background] Chihara G, Maeda Y, Hamuro J, Sasaki T, Fukuoka F. Inhibition of mouse sarcoma 180 by polysaccharides from Lentinus edodes (Berk.) sing. Nature. 1969 May 17;222(5194):687-8. doi: 10.1038/222687a0. No abstract available. PMID 5768289
- See also: Meiji University of Oriental Medicine — http://www.meiji-u.ac.jp/